CLINICAL TRIAL: NCT06354127
Title: A Multi-center, Randomized, Double-blind, Positive Drug-controlled Clinical Study to Evaluate the Safety and Efficacy of Botulinum Toxin Type A for Injection in the Treatment of Moderate to Severe Glabellar Lines
Brief Title: DWP450 for Treating Moderate to Severe Glabellar Lines
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Daewoong Pharmaceutical Co. LTD. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DW_DWP450009
Record Dates: First submitted 2024-04-03; First posted 2024-04-09 (Actual); Last update posted 2024-04-09 (Actual); Status verified 2024-04

CONDITIONS: Moderate to Severe Glabellar Lines
MeSH Terms: interventions — DWP450; Botulinum Toxins, Type A

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DWP450 (Experimental)
  Interventions: Drug: DWP450
- Botox® (Active Comparator)
  Interventions: Drug: Botox®

INTERVENTIONS:
Drug: DWP450 — The test drug or control drug is injected on the day of administration.
  Arms: DWP450
Drug: Botox® — The test drug or control drug is injected on the day of administration.
  Arms: Botox®

SUMMARY:
A multi-center, randomized, double-blind, positive drug-controlled clinical study to evaluate the safety and efficacy of Botulinum Toxin Type A for Injection in the treatment of moderate to severe glabellar lines

ELIGIBILITY:
Inclusion Criteria:

* Adult males or females aged 20-65 years old.
* Moderate to severe (grade 2-3) glabellar lines based on investigator's assessment of severity of glabellar lines at maximum frown.

Exclusion Criteria:

* Having received any glabellar (including forehead) cosmetic procedures/surgeries, such as dermal filling, face lifting, photoelectric therapy, hydro lifting, microneedle, chemical peeling or scar removal surgery, or dermabrasion within 6 months prior to screening.
* Planning to receive any facial cosmetic procedures/surgeries, including but not limited dermal filling, face lifting, photoelectric therapy, hydro lifting, microneedle, chemical peeling or scar removal surgery, during the study period.
* Skin infection at injection site or systemic skin disease assessed with the potential to interfere with efficacy evaluation or safety evaluation of glabellar lines or forehead lines.
* Glabellar lines that cannot be fully flattened through surgery, by hand or by other methods.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 473 (Actual)
Dates: Start 2020-08-12 (Actual); Primary Completion 2020-11-24 (Actual); Study Completion 2021-01-25 (Actual)

PRIMARY OUTCOMES:
Response rate based on the investigator's on-site assessment of severity of glabellar lines at maximum frown | Week 4
  The difference between the two groups in response rate at Week 4 based on the investigator's on-site assessment of severity of glabellar lines (at maximum frown).

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Ninth People's Hospital, Shanghai Jiaotong University School of Medicine, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No